CLINICAL TRIAL: NCT04727632
Title: [18F]Fluoroestradiol-PET/CT Companion Imaging Study to the FORESEE: Functional Precision Oncology for Metastatic Breast Cancer Feasibility Trial
Brief Title: [18F]Fluoroestradiol-PET/CT Companion Imaging Study to the FORESEE Trial
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: It was not feasible to perform FES PET/CT
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI140278
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Estrogen Receptor Positive Breast Cancer
MeSH Terms: interventions — proto-oncogene protein c-fes-fps

STUDY DESIGN:
Intervention Model Description: This is a companion imaging study to IRB # 131027 FORESEE: Functional precision oncology for metastatic breast cancer: a feasibility trial. This companion imaging study will obtain [18F]Fluoroestradiol (FES)-PET/CT imaging of breast cancer patients refractory to all combinatorial hormonal therapies enrolled in the FORESEE trial and correlate the FES-PET/CT results with data from FORESEE including estrogen receptor (ER) status and drug profiling results from patient-derived organoid models.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: all patients (Experimental): One session of [18F]FES PET/CT Imaging
  Interventions: Drug: [18F]Fluoroestradiol (FES) PET/CT

INTERVENTIONS:
Drug: [18F]Fluoroestradiol (FES) PET/CT — [18F]Fluoroestradiol (FES) PET/CT

SUMMARY:
This protocol is a companion imaging study that will add FES-PET/CT imaging to the FORESEE trial at HCI. This study will establish the feasibility of using FES-PET/CT imaging to guide therapeutic decision making for functional precision oncology trials. The unique ability of FES-PET/CT to show absence of functional estrogen receptors throughout the entire body may improve confidence among research oncologists that an ER+ metastatic breast cancer patient is truly refractory to hormonal therapies which is a critical determination in the study design of the FORESEE trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or greater.
* All patients or legal guardians are willing and able to sign written informed consent and HIPAA authorization in accordance with local and institutional guidelines.
* Enrolled on the FORESEE trial.
* Biopsy proven estrogen receptor positive breast cancer.
* Patient deemed refractory to all combinations of hormonal therapies by FORESEE trial investigators.

Exclusion Criteria:

* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals. Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion.
* Patients who require monitored anesthesia for PET/CT scanning.
* Patients who are too claustrophobic to undergo PET/CT scanning.
* Patients who are pregnant or currently breast feeding.
* Any patient that is medically unstable defined as a patient requiring inpatient hospitalization or needing evaluation at an acute care or urgent care facility at the time of imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Number of patients on the FORESEE trial refractory to all combinatorial hormonal therapies that are recruited and imaged with FES-PET/CT prior to switching to non-hormonal therapeutic agents | 12 weeks
  establish proof-of-concept to inform use of FES-PET/CT in future larger precision oncology trials

SECONDARY OUTCOMES:
Rate of concordance between FES-PET/CT imaging (positive or negative uptake) and ER status from tumor biopsy | 12 weeks
  assess FES-PET/CT concordance with ER status from patient-derived organoid models and concordance between FES-PET/CT imaging and patient-derived organoid drug profiling results for predicting response to hormonal therapies
Rate of concordance between positive FES-PET/CT scan and response to hormonal therapies from drug profiling results using patient-derived organoid models | 12 weeks
  assess FES-PET/CT concordance with ER status from patient-derived organoid models and concordance between FES-PET/CT imaging and patient-derived organoid drug profiling results for predicting response to hormonal therapies

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Covington, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No